CLINICAL TRIAL: NCT06302101
Title: Efficacy of Synchronous Telerehabilitation Chair-Based Exercises and Cognitive Exercises in Elderly Individuals
Brief Title: Telerehabilitation Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, Assistant Professor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise in older adults
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-05

CONDITIONS: Pain; Elderly; Balance
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- İntervention (Experimental): chair-based exercises and cognitive exercises
  Interventions: Behavioral: chair-based exercises; Behavioral: cognitive exercises
- Control group (Active Comparator): chair-based exercises
  Interventions: Behavioral: chair-based exercises

INTERVENTIONS:
Behavioral: chair-based exercises — Synchronous online telerehabilitation chair-based exercises will be performed under the supervision of a physiotherapist twice a week for 8 weeks for intervention group.
  The control group will be given a brochure with explanations of the exercises.
Behavioral: cognitive exercises — Cognitive exercises will be performed under the supervision of a physiotherapist 1 day a week for 8 weeks as online telerehabilitation for intervention group.
  Arms: İntervention

SUMMARY:
The aim of this study was to investigate the effectiveness of chair-based exercises and cognitive exercises through synchronous telerehabilitation in older adults.

Older adults will be divided into two groups (intervention group n=16; control group n=11) .

ELIGIBILITY:
Inclusion Criteria:

* Getting a score of 6 or above on the Hodkinson Mental Test

Exclusion Criteria:

* -Having another chronic disease that can cause pain Having a neurological disease Being blind Having an orthopedic, neurological or mental disability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 15 minutes
  It is a scale consisting of 14 items.The maximum score is 56.
Timed Up and Go Test During Dual Tasking | 5 minutes
  While performing the timed up and go test, the person will be asked to count backwards from 100, two by two.
Geriatric Pain Measure | 15 minutes
  It is a multidimensional scale with 24 items.Scores range from 0-100.
Older people's quality of life-brief (OPQOL-brief) | 8 minutes
  It consists of 13 items. Scores between 13 and 65 can be obtained, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Hodkinson Mental Test | 5 minutes
  The test consists of 10 questions in total.total score is between 0-10
Dominant Side One Leg Stand Test | 30 seconds
  The dominant leg will be asked to lift up. The time will end when the foot touches the ground.
Timed Up and Go Test | 3 minutes
  An area of 3 meters will be determined. The individual will be asked to get up from the chair, walk, come back and sit down without any support.
chair sit and stand test | 30 seconds
  You will be asked to stand up and sit down quickly for 30 seconds
Geriatric Depression Scale | 15 minutes
  It consists of 30 items. A score between 0-15 is received.
Successful Aging Scale | 5 minutes
  It consists of ten questions.A minimum of 10 and a maximum of 70 points can be obtained from this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Gur Kabul, Uşak, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kabul EG, Akar B, Calik BB. Effectiveness of Chair-Based Exercises and Cognitive Training With Synchronous Telerehabilitation Method in Healthy Older Adults: A Pilot Randomised Controlled Study. Psychogeriatrics. 2025 Nov;25(6):e70100. doi: 10.1111/psyg.70100. PMID 40983490